CLINICAL TRIAL: NCT02259257
Title: 3D/4D Ultrasound Contrast Enhanced Imaging (CEUS) for Carotid Plaque Vulnerability
Acronym: CEUS carotid
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Diana Gaitini MD. (Other)
Collaborators: Technion, Israel Institute of Technology (Other); Rush University (Other)
Responsible Party: Sponsor-Investigator, Diana Gaitini MD., Director Ultrasound Unit, Dept of Medical Imaging, Rambam Health Care Campus
Organization: Rambam Health Care Campus (Other)
Other Study IDs: 226-14 RMB CTIL
Record Dates: First submitted 2014-09-23; First posted 2014-10-08 (Estimated); Last update posted 2014-10-08 (Estimated); Status verified 2014-10

CONDITIONS: Atherosclerosis; Stroke
Keywords: carotid arteriosclerosis; contrast-enhanced ultrasound; neovascularization; quantitative analysis; 3D/4D imaging; CEUS; Vasa vasorum
MeSH Terms: conditions — Atherosclerosis; Stroke; Carotid Artery Diseases; Neovascularization, Pathologic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue: Carotid plaque histological specimen
Oversight: Data Monitoring Committee: No

SUMMARY:
Contrast enhanced 3D/4D (3 dimension/4 dimension) ultrasound (CEUS) provides visualization of the dynamic vascular features of the plaques, in a unique spatial format using three orthogonal planes and angiogram-like images. Therefore, the observer can utilize the entire vascular system in a volumetric manner (3D). The rotation of the intra-plaque neovasculature as viewed in various angles provides a realistic representation that is more easily appreciated. Inter-observer variability for individual plaques has been assessed and inter-observer variability and inter-scan variability (the analysis of multiple images from single patients in longitudinal studies) were dependent on plaque size, with larger plaques showing lower variability. Therefore, the proposed 3D/4D vs. 2D CEUS imaging of the carotid plaque will provide added value for the depiction of the and quantification of intra-plaque blood vessel density by providing a true volumetric viewing area. This data will be correlated to the subsequent surgical specimens. The goal of the protocol is to investigate the correlation of intra-plaque blood vessel density and hemorrhage to 3D/4D CEUS vasa vasorum using quantitative software analyses. The histology methods used for quantification of hemorrhage and vessel density analyses.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects with known carotid artery disease will be included.
* Subject must be able and willing to comply with study procedures and provide a signed and dated informed consent including consent for 3 year annual follow up.
* Subjects will be screened by asking each study subject if they have known or suspected hypersensitivity to any of the components of Optison, blood, blood products of albumin. In addition, each study subject will be asked if they have a right to left or bi-directional or transient right to left cardiac shunts. If any of the above questions are answered in the positive, the patient will not be eligible for inclusion in the study.

Exclusion Criteria:

* Female subjects of child bearing potential will be excluded.
* The subject presents any clinically active, serious, life-threatening disease, with a life expectancy of less than 1 month or where study participation may compromise the management of the subject or other reason that in the judgment of the investigator makes the subject unsuitable for participation in the study.
* History of acute occlusion requiring medical intervention of any artery (including aorta) within 6 months of consent.
* Has a known or suspected hypersensitivity to any of the components of Optison, blood, blood products, or albumin.
* Has known right to left, bi-directional or transient right to left cardiac shunts.
* Any known contra-indications as listed on the current Optison package insert.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for endarterectomy due to carotid stenosis demonstrated on a previous imaging examination (exhibiting >50% intra-luminal narrowing or a maximum IMT measurement of > 1.5mm) or have experienced a CVA event (TIA/CVA) .
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Carotid plaque vascularization as seen on CEUS and histology compared to 3 year follow up of cardiovascular events. | Post processing of CEUS will be done up to 3 years post surgery
  Post processing of CEUS data for carotid plaque vascularization.
  In addition all carotid artery histology specimens, routinely obtained at the time of surgery at each center, will be analyzed to include the following tissue stains: CD3, CD31, CD38 and Hemosiderin.

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Health Care Center, Haifa, Haifa District, Israel

REFERENCES:
- [Background] Hoogi A, Adam D, Hoffman A, Kerner H, Reisner S, Gaitini D. Carotid plaque vulnerability: quantification of neovascularization on contrast-enhanced ultrasound with histopathologic correlation. AJR Am J Roentgenol. 2011 Feb;196(2):431-6. doi: 10.2214/AJR.10.4522. PMID 21257897
- [Background] Staub D, Schinkel AF, Coll B, Coli S, van der Steen AF, Reed JD, Krueger C, Thomenius KE, Adam D, Sijbrands EJ, ten Cate FJ, Feinstein SB. Contrast-enhanced ultrasound imaging of the vasa vasorum: from early atherosclerosis to the identification of unstable plaques. JACC Cardiovasc Imaging. 2010 Jul;3(7):761-71. doi: 10.1016/j.jcmg.2010.02.007. PMID 20633855
- [Background] Michel JB, Virmani R, Arbustini E, Pasterkamp G. Intraplaque haemorrhages as the trigger of plaque vulnerability. Eur Heart J. 2011 Aug;32(16):1977-85, 1985a, 1985b, 1985c. doi: 10.1093/eurheartj/ehr054. Epub 2011 Mar 12. PMID 21398643
- [Background] Hellings WE, Peeters W, Moll FL, Piers SR, van Setten J, Van der Spek PJ, de Vries JP, Seldenrijk KA, De Bruin PC, Vink A, Velema E, de Kleijn DP, Pasterkamp G. Composition of carotid atherosclerotic plaque is associated with cardiovascular outcome: a prognostic study. Circulation. 2010 May 4;121(17):1941-50. doi: 10.1161/CIRCULATIONAHA.109.887497. Epub 2010 Apr 19. PMID 20404256
- [Background] Sluimer JC, Daemen MJ. Novel concepts in atherogenesis: angiogenesis and hypoxia in atherosclerosis. J Pathol. 2009 May;218(1):7-29. doi: 10.1002/path.2518. PMID 19309025
- [Background] Shah F, Balan P, Weinberg M, Reddy V, Neems R, Feinstein M, Dainauskas J, Meyer P, Goldin M, Feinstein SB. Contrast-enhanced ultrasound imaging of atherosclerotic carotid plaque neovascularization: a new surrogate marker of atherosclerosis? Vasc Med. 2007 Nov;12(4):291-7. doi: 10.1177/1358863X07083363. PMID 18048465